CLINICAL TRIAL: NCT00820521
Title: Ascending Single Dose Study of the Safety, Tolerability, and Pharmacokinetics of GAP-134 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating Single Doses of GAP-134
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 3205A2-1003
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- active (Experimental)
  Interventions: Drug: active
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: active
  Arms: active
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ascending single oral doses of GAP-134 in healthy subjects, to provide the initial pharmacokinetic profile of the oral formulation of GAP-134 in healthy subjects, and to evaluate the effect on the pharmacokinetic profile of a high-fat meal of 450 mg of GAP-134 administered to healthy subjects.

ELIGIBILITY:
Inclusion Criteria

* Men or women of nonchildbearing potential (WONCBP) aged 18 to 50 years inclusive at screening.
* WONCBP may be included if they are either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for ≥1 year (with follicle stimulating hormone [FSH] level ≥38 mIU/mL) and must have a negative pregnancy test result within 24 hours before administration of the study drug or placebo.
* Women who are surgically sterile must provide documentation of the procedure by an operative report or by an ultrasound scan report.
* Sexually active men must agree to use a medically acceptable form of contraception during the study and continue using it for 12 weeks after study drug or placebo administration.
* Body mass index (BMI) in the range of 18.0 to 30.0 kg/m2 and body weight ≥50 kg.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital sign measurements, and 12-lead electrocardiogram (ECG).
* Serum creatinine level must be less than 1.30 mg/dL. (Normal range: 0.44 to 1.24 mg/dL.)
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.

Exclusion Criteria

* Presence or history of any disorder that may prevent the successful completion of the study.
* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the study drug or placebo.
* Acute disease state (eg, nausea, vomiting, fever, or diarrhea) within 7 days before administration of study drug or placebo.
* Any history of clinically important cardiac arrhythmias.
* Familial history of long QT syndrome or unexpected cardiac death.
* History of drug abuse within 1 year before before administration of study drug or placebo.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability will be evaluated from reported AEs, scheduled physical examinations, vital sign measurements, cardiac rhythm monitoring, 12 lead ECGs, and clinical laboratory test results. | 2 months

SECONDARY OUTCOMES:
pharmacokinetic parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer